CLINICAL TRIAL: NCT06032260
Title: The Effects of a Fiber-enriched Bakery Product on Glucose, Insulin Values and Appetite. A Pilot Randomized Cross-over Trial
Brief Title: The Effects of a Fiber-enriched Bakery Product on Glucose, Insulin Values and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: PAN_2023
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Arabinoxylan; fiber-enriched product; glycemia; insulin; appetite
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: crossover randomized double-blind trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the participant nor the investigators were aware of the composition of the administered food. The two types of foods were identical for packages, color, flavor, smell, and appearance. Furthermore, the researchers who analyzed data and the laboratory personnel who performed the biochemical analyses were blinded to the group assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enriched panettone (Experimental): 100 grams of panettone enriched with fiber. The added fiber is JAX Plus® (Heallo srl, Milano, Italy), a soluble fiber with Arabinoxylans from wheat and barley
  Interventions: Other: Enriched panettone
- Panettone standard (Active Comparator): 100 grams of panettone without fiber enrichment
  Interventions: Other: Panettone standard

INTERVENTIONS:
Other: Enriched panettone — Volunteers consumed 100 grams of panettone enriched with fiber (JAX Plus® (Heallo srl, Milano, Italy), a soluble fiber with Arabinoxylans from wheat and barley
  Arms: Enriched panettone
Other: Panettone standard — Volunteers consumed 100 grams of panettone standard
  Arms: Panettone standard

SUMMARY:
The aim of the present pilot randomized controlled trial is to compare the effects of the following: 1)-panettone enriched with arabinoxylans (p-rich), 2)-panettone not enriched (p-standard) on blood glucose and insulin values, and appetite scores in 10 healthy volunteers.

DETAILED DESCRIPTION:
This is a crossover, randomized double-blind trial. A product enriched with arabinoxylan extracted from threshing (panettone, p-rich, a sweet baked product with a high glycemic index) was developed to assess the impact on metabolic responses and satiety when compared to the standard product (p-standard) .

Ten Caucasian non-smoker healthy adult volunteers were enrolled starting from January 2023.

Participants were randomized to receive either the p-rich or p-standard. The order of administration of each product was randomized using a computer-generated sequence. The day of each test, fasting individuals underwent a blood sample collection, and weight and height measurements. Then, participants consumed 100 grams of the product within 20 minutes, while sitting. Blood samples were collected at 15, 30, 45, 60, 90, 120 minutes after the consumption of each food.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers healthy adults;
* age 20-65 years;
* ability to provide informed written consent

Exclusion Criteria:

* obesity;
* chronic diseases or pharmacological therapies;
* dietary restrictions;
* allergy or intolerance to the tested food

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in circulating concentrations of glucose | 15, 30, 45, 60, 90, 120 minutes after the consumption of each food
  To evaluate changes in glucose responses after the consumption of p-rich when compared to p-standard

SECONDARY OUTCOMES:
Changes in circulating concentrations of insulin | 15, 30, 45, 60, 90, 120 minutes after the consumption of each food
  To evaluate changes in insulin responses after the consumption of p-rich when compared to p-standard
Changes in subjective appetite score (VAS) | 60, 120, 180, and 240 minutes after the consumption of each food
  To evaluate changes in appetite responses after the consumption of p-rich when compared to p-standard. Subjective sensations of appetite were assessed by a visual analogue scale (VAS) ranging from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, AT, Italy

IPD SHARING:
Plan to Share IPD: No